CLINICAL TRIAL: NCT05360823
Title: The Effect of Using a Birth Ball and Squatting Position During Labor on Labor Pain, Duration of Labor and Satisfaction
Brief Title: The Effect of Using a Birth Ball and Squatting Position During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Dünmez (Other)
Responsible Party: Sponsor-Investigator, Fatma Dünmez, Midwifery-Master Student, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ISBASP
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Labor Pain; Labor Fast; Satisfaction, Patient
Keywords: Labor Pain; Birth ball; Squatting; Duration of labor; Satisfaction
MeSH Terms: conditions — Labor Pain; Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Birth Ball Group (Experimental): In the active and transitional phases, during contractions, performing exercises on the birth ball (fully rotating the hip, moving to the right/left, coming back and forth, and slightly bouncing while sitting on the birth ball) (average 25 minutes). In order to monitor the condition of the fetus, exercises on the birth ball were performed by the pregnant woman during contractions while connected to NST.
  Interventions: Other: Birth ball
- Squatting Group (Experimental): In the active and transitional phase, squatting position (squatting with feet shoulder-width apart by laying a clean sheet on the floor and getting support from a bed, chair or birth ball) during contractions (average 25 minutes). In order to monitor the condition of the fetus, the squatting position was used by the pregnant woman during contractions while connected to the NST.
  Interventions: Other: Squatting
- Control Group (No Intervention): Usual routine care of the service.

INTERVENTIONS:
Other: Birth ball — Exercises for childbirth
  Arms: Birth Ball Group
Other: Squatting — Exercises for childbirth
  Arms: Squatting Group

SUMMARY:
The aim of the study was to evaluate the effect of using the birth ball and squatting position during labor on labor pain, duration of labor and satisfaction. The research is a randomized controlled experimental study. The sample of the study consisted of a total of 159 pregnant women, 53 in the birthing ball application group, 53 in the squatting group, and 53 in the control group, who met the criteria for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* No risky pregnancy
* Gestational week between 37-42
* Unopened amniotic membrane
* Those who will give birth vaginally
* In active phase
* Fluent in Turkish
* Singleton pregnancy
* Primiparous

Exclusion Criteria:

* Any complication development
* Cesarean section status

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Personal and Obstetric Information Form | pre-intervention
  This form, prepared by the researcher, consists of 45 questions including sociodemographic, obstetric and obstetric follow-up information of women.
Visual Analog Scale (VAS) | latent, active and transition phase of labor
  It is a measuring instrument with a score between 0 (no pain) and 10 (severe pain), divided equally by marks on a horizontal or vertical 10 cm line. Horizontal form was used in the research. The scale was used to assess the severity of pain.
Partogram | active phase of labor
  It is a graphical form used to evaluate the progress of birth and the health status of the baby.
Evaluation Scale for Maternal Satisfaction with Normal Delivery | Postpartum at the 4th hour
  This is used to assess the mother's level of satisfaction at birth. The scale, which has a validity and reliability of 0.91 in Turkey, was developed by Güngör and Beji in 2009. It is a 5-point Likert-type scale consisting of 43 items and 10 sub-dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Dünmez, Midwife, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Yeung MPS, Tsang KWK, Yip BHK, Tam WH, Ip WY, Hau FWL, Wong MKW, Ng JWY, Liu SH, Chan SSW, Law CK, Wong SYS. Birth ball for pregnant women in labour research protocol: a multi-centre randomised controlled trial. BMC Pregnancy Childbirth. 2019 May 6;19(1):153. doi: 10.1186/s12884-019-2305-8. PMID 31060522
- [Background] Lavender T, Cuthbert A, Smyth RM. Effect of partograph use on outcomes for women in spontaneous labour at term and their babies. Cochrane Database Syst Rev. 2018 Aug 6;8(8):CD005461. doi: 10.1002/14651858.CD005461.pub5. PMID 30080256
- [Background] Gungor I, Beji NK. Development and psychometric testing of the scales for measuring maternal satisfaction in normal and caesarean birth. Midwifery. 2012 Jun;28(3):348-57. doi: 10.1016/j.midw.2011.03.009. Epub 2011 May 4. PMID 21546142
- [Derived] Dunmez F, Yilmaz T. The effect of using birth ball and squatting position during labor on pain, duration, and satisfaction: A randomized controlled trial. Jpn J Nurs Sci. 2024 Apr;21(2):e12580. doi: 10.1111/jjns.12580. Epub 2023 Dec 10. PMID 38073180
- See also: Ministry of Health Partograph Circular — https://shgmkalitedb.saglik.gov.tr/Eklenti/6486/0/partografgenelgesipdf.pdf